CLINICAL TRIAL: NCT01542203
Title: Impact of Body Weight on the Pharmacokinetic Analysis of Doxorubicin and Cyclophosphamide in Breast Cancer Patients
Brief Title: Impact of Body Weight on Pharmacokinetic Analysis of Doxorubicin + Cyclophosphamide in Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: study is classified as ancillary / correlative
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 062011-056
Record Dates: First submitted 2012-02-20; First posted 2012-03-02 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: doxorubicin; cyclophosphamide; Breast Cancer; BMI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer, Various BMIs: 18 female breast cancer patients who are normal weight (body mass index [BMI] < 25 kg/m2, overweight or class I obese(BMI 25-34.9 kg/m2), or class II-III obese (BMI > 35 kg/m2).

SUMMARY:
This single site study will be conducted at the UT Southwestern Simmons Cancer Center. This study is designed to measure drug concentrations in the blood of 18 female breast cancer patients who require doxorubicin (30 minute infusion) and cyclophosphamide (30 minute infusion) as part of standard medical care. Up to a total of 40 adult female participants will be consented for the study at the cancer center. Eighteen of these participants are needed to complete the study. The others will likely be screen failures. The participants will have no more than 100 ml of blood drawn via a peripheral intravenous catheter just prior to the doxorubicin infusion, and then at 0.5, 1, 1.5, 2, 3, 4, 5, 12-24, and 24-72 h after the beginning of the doxorubicin infusion. The 5 hour blood draw is optional. The intravenous catheter will be removed when the participant is discharged from the cancer center on day 1. The participant will be asked to return to the cancer center at 12-24 and 24-72 hours to have the final 2 blood draws conducted. The participants must be treated with Doxorubicin and Cyclophosphamide in order to participate in this pharmacokinetic analysis study.

DETAILED DESCRIPTION:
The study will require a total of 11 participant contacts over 3 days (1 day outpatient clinic visit for doxorubicin and cyclophosphamide infusions and blood draws, 2 follow up outpatient clinic visits for blood draws) with no more than 100 mL of blood being drawn. All blood draws will be collected for the purpose of research.

Screening and Informed Consent Procedures

1. The participant's height, weight, medical history, comorbid conditions, and current medications will be obtained from the electronic medical record (EMR).

   Update 1 : January 12, 2012
2. Study personnel will provide the participant with additional information about the study and provide the participant with the opportunity to ask any questions. Each participant will then be asked if she is willing to provide informed consent.
3. Information from the routine physical examination including vital signs (temperature,respiratory rate, blood pressure, heart rate) will be collected from the medical chart.

Procedures and Evaluation during the Research

1. Each participant will then have no more than10ml of blood drawn 8 times, at t=0h (predose),at the end of the doxorubicin infusion, at the end cyclophosphamide infusion, and 1.5, 2, 3, 4, 5, 12-24, and 24-72 h following the beginning of doxorubicin infusion. All blood draws will be performed using the peripheral intravenous catheter being used for standard medical care. Labels on blood samples will not contain participant name, but a randomly generated participant identification number.
2. All blood samples will placed on ice and immediately transported to Dr. Richard Leff's laboratory for sample preparation.9 Samples will be spun in a refrigerated centrifuge and then placed in a -80oC freezer. As explained below, Dr. Leff or his laboratory will not have access to any participant identifiers.
3. The participant is discharged from the cancer center (for research purposes) after the 4 hour blood draw, unless the participant is willing to stay for the 5 hour blood draw.
4. The participant will return to the cancer center at 12-24 and 24-72 hours for blood draws.
5. The participant is discharged from the study after the 24-72h blood draw. Follow-up: Participants will be asked to return to the cancer center for 12-24 and 24-72 hour blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Females,
* age 18 years of age or older, of all racial and ethnic origins that are scheduled to receive the first cycle of a single intravenous dose of doxorubicin (30 minute infusion) and cyclophosphamide (30 minute infusion) as part of standard medical care for breast cancer.
* English and/or Spanish speaking participants are eligible to participate.

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of doxorubicin and cyclophosphamide on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of doxorubicin or cyclophosphamide, so that the pregnancy and post-partum state would be a confounding variable.
* Participants unwilling to comply with study procedures.
* CrCl < 10 ml/min
* Participants requiring peritoneal or hemodialysis
* Serum bilirubin > 1.19 mg/dL
* Receipt of the following drugs that:

  * Alter doxorubicin concentrations: carbamazepine, cyclosporine, fosphenytoin, paclitaxel, phenytoin, sorafenib, valspodar, verapamil
  * Alter cyclophosphamide concentrations: cyclosporine, nevirapine, ondansetron
  * All other drugs will be reviewed during screening of the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06-25 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UTSouthwestern Medical Center, Dallas, Texas, United States